CLINICAL TRIAL: NCT04199247
Title: Initiation of an Early Exercise Program to Improve Symptoms and Psychosocial Function After Pediatric Mild Traumatic Brain Injury
Brief Title: Early Exercise to Improve Psychosocial Function After Pediatric Mild Traumatic Brain Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-2020
Record Dates: First submitted 2019-12-10; First posted 2019-12-13 (Actual); Last update posted 2022-05-04 (Actual); Status verified 2022-05

CONDITIONS: Brain Concussion; Pediatric; Mild Traumatic Brain Injury; Psychological
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Intervention Model Description: Within 1 week of injury, participants will be randomized to either a sub symptom threshold exercise program (intervention group) or usual care (recommendation from their doctor). Those in the intervention group will participate in an exercise program 5x/week, 20-30 minutes/session, for 2 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise (Experimental): Within 1 week of injury, participants will be randomized to either a sub symptom threshold exercise program (intervention group) or usual care (recommendation from their doctor). Those in the intervention group will participate in an exercise program 5x/week, 20-30 minutes/session, for 2 months.
  Interventions: Behavioral: Sub symptom aerobic exercise
- Usual Care (No Intervention): Participants will continue with their return to play progression based upon the advice given to them at their initial post-injury evaluation.

INTERVENTIONS:
Behavioral: Sub symptom aerobic exercise — Participants will meet with a member of the research team to undergo a bike-based exercise test at the initial test. Heart rate will be obtained at the completion of the test, and intervention participants will be asked to complete exercise at 80% of that level, 5x/week for 20-30 minutes/session over the next two months.
  Arms: Exercise

SUMMARY:
The investigators will test the central hypotheses according to the following Specific Aims:

Aim 1. Determine if an individually prescribed exercise program initiated within the first week of mild traumatic brain injury can reduce the risk of developing persistent post-concussion symptoms relative to usual care. The investigators hypothesize that the exercise group will have a lower risk of developing persistent post-concussion symptoms than the usual care group.

Aim 2. Examine the effect of a two-month exercise program on psycho-social, pain interference, and sleep outcomes following mild traumatic brain injury. The investigators hypothesize the exercise group will report lower anxiety, depression, and pain interference ratings, and higher peer relationship and sleep quality ratings two months of exercise following mild traumatic brain injury compared to usual care.

DETAILED DESCRIPTION:
The long-term research goal of the proposed study is to develop individualized sub-symptom exercise prescriptions for youth who sustain mild traumatic brain injury that can help to alleviate mild traumatic brain injury symptoms, reduce the risk of persistent post-concussion symptoms, and improve psychosocial outcomes. The overall objectives of this application are to prospectively (1) determine if a prescribed exercise program initiated within the first week of mild traumatic brain injury can reduce the risk of developing persistent post-concussion symptoms and (2) examine the effects of an exercise program on psychosocial, sleep, and pain outcomes when initiated within 7 days of injury and continued for two months. The investigators will address these objectives by testing the central hypotheses that those assigned to an exercise intervention will have lower risk of developing persistent post-concussion symptoms and will report lower anxiety, depression, and pain interference ratings, higher peer relationship ratings, and better sleep quality ratings compared to usual care. In order to achieve this, the investigators will use a block stratified randomized intervention design. Block stratified randomization procedures will be conducted according to standard procedures so that sample numbers are equally assigned to each group, selected due to the relatively small sample size of the proposed study. Participants will be identified, enrolled, and assessed within 5 days of mild traumatic brain injury, randomized to an exercise intervention or usual care group 3-7 days after mild traumatic brain injury, and follow-up with in person assessments at approximately one and two months post-injury.

ELIGIBILITY:
Inclusion Criteria:

1. Concussion or mTBI diagnosis by a board-certified Sports Medicine physician, pediatric Emergency Medicine physician, general pediatrician physician, or advanced practice provider under the direction of a physician. This will be defined in a similar manner according to available guidelines: a direct or indirect blow to the head, face, neck, or elsewhere that manifests with the presence of symptoms and neurological impairment
2. Aged 10 - 18 years to ensure a pediatric sample of participants.
3. A persistent postconcussion symptom risk score ≥ 9 to ensure all participants are in the high risk of persistent postconcussion symptom category.
4. A Post-Concussion Symptom Inventory score > 9 to ensure participants have not recovered by the time they enroll in the study.
5. Access to an internet connection (via computer or smart phone) so that physical activity and exercise can be tracked via heart rate monitor.

Exclusion Criteria:

1. Concurrent lower extremity injury so that exercise testing results are not confounded by other injury.
2. Aerobic exercise contraindication so that participants are able to complete the exercise testing protocol.
3. Diagnosed mild traumatic brain injury by a healthcare provider within 6 months of qualifying injury to ensure that residual effects of prior mild traumatic brain injury do not bias the results of our investigation.
4. Mild traumatic brain injury that results in positive findings on neuroimaging, or extra-axial or intraparenchymal bleeds to avoid potential injuries that are more severe than mild traumatic brain injury.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2020-02-20 (Actual); Primary Completion 2021-11-08 (Actual); Study Completion 2021-11-08 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in Post Concussion Symptom Inventory | Baseline (within 1 week of injury), Month 1, Month 2
  Overall symptom severity, rated as a sum score from 0-122. A higher score indicates more severe symptoms, while a 0 indicates that the patient is not experiencing symptoms.

SECONDARY OUTCOMES:
Change from Baseline in Patient-Reported Outcomes Measurement Information System (PROMIS) Short Form Pediatric 25 | Baseline (within 1 week of injury), Month 1, Month 2
  A brief generalized quality of life questionnaire. We will calculate the sub-scale scores for the domains of Mobility, Depressive Symptoms, Anxiety, Peer Relationships, and Pain Interference. Each sub-scale is calculated as a sum of 4 questions, rated from 0-4. Thus, each subscale is from 0-16, where a 16 indicates a greater presence of the domain being measured.
Change from Baseline in Tampa Scale of Kinesiophobia | Baseline (within 1 week of injury), Month 1, Month 2
  A brief questionnaire about fear of movement and injury related to returning to sport. The subject answers 18 questions rated from 1 (strongly disagree) to 4 (strongly agree). There is a total sum score ranging form 18-72, where a higher score represents more fear of movement.
Change from Baseline in Physical activity level | Baseline (within 1 week of injury), Month 1, Month 2
  In order to assess the effect of physical activity level on recovery, we will provide participants with heart-rate activity monitors.
Change from Baseline in Dual-task walking speed | Baseline (within 1 week of injury), Month 1, Month 2
  Measure of the the average walking speed of subjects during dual-task conditions (m/s).

CONTACTS AND LOCATIONS:
Overall Officials: David R Howell, PhD, Principal Investigator — Children's Hospital Colorado
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No